CLINICAL TRIAL: NCT06391853
Title: Investigating Brain Insulin Resistance in Alzheimer Disease with Intra-Nasal Insulin Administration: a Multimodal Neuroimaging Study
Brief Title: Investigating Brain Insulin Resistance in Alzheimer Disease with IntraNasal Insulin : a Multimodal Neuroimaging Study
Acronym: Memori³
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not realisable on time planned and with the academic funds
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SRB2023-183; 2023-508203-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-08; First posted 2024-04-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Intranasal Insulin
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intranasal Insulin then Placebo (Experimental): First day , participant will receive Intranasal Insulin (100IU insulin/ml) 2 spray representing 0.8 ml in each nostril to achieve 1.6 ml (total dose =160UI)
  Second day participant will receive Placebo Intranasal , witch is saline solution (Nacl 0.9%). 2 spray representing 0.8 ml in each nostril to achieve 1.6 ml
  Interventions: Drug: Insulin
- Placebo then Intranasal Insulin (Active Comparator): First day ,participant will receive Placebo Intranasal , witch is saline solution (Nacl 0.9%). 2 spray representing 0.8 ml in each nostril to achieve 1.6 ml
  Second day, participant will receive Intranasal Insulin (100IU insulin/ml) 2 spray representing 0.8 ml in each nostril to achieve 1.6 ml (total dose =160UI)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin — A venous line will be installed and an MRI-compatible EEG Cap (32 scalp electrodes) will be installed with conductive gel between the scalp and the electrode.
  Participants will receive 2 Intranasal spray. Participants will then be installed in the PET/MRI camera. At 30 min post INI administration, a continuous infusion of FDG will be started, along with dynamic PET acquisition while recording EEG and fMRI sequences. Participant will be asked to rest, eyes opened and awake to stay awake during the 55 minutes.
  At the end of the neuroimaging data acquisition, participants will be freed from EEG Cap and will undergo neuropsychologic evaluation.The final part of neuropsychological evaluation will be performed on week later, on the phone.. The total study time for each scanning day will be around 3h.
  Other Names: FDG-PET; EEG; fMRI
  Arms: Intranasal Insulin then Placebo
Drug: Placebo — A venous line will be installed and an MRI-compatible EEG Cap (32 scalp electrodes) will be installed with conductive gel between the scalp and the electrode.
  Participants will receive 2 Intranasal spray. Participants will then be installed in the PET/MRI camera. At 30 min post INI administration, a continuous infusion of FDG will be started, along with dynamic PET acquisition while recording EEG and fMRI sequences. Participant will be asked to rest, eyes opened and awake to stay awake during the 55 minutes.
  At the end of the neuroimaging data acquisition, participants will be freed from EEG Cap and will undergo neuropsychologic evaluation.The final part of neuropsychological evaluation will be performed on week later, on the phone.. The total study time for each scanning day will be around 3h.
  Other Names: FDG-PET; EEG; fMRI
  Arms: Placebo then Intranasal Insulin

SUMMARY:
Using simultaneous multimodal neuroimaging (FDG-PET, fMRI, EEG), this research project will aim to further investigate in vivo brain insulin signalling by exploring the effects of acute INI administration on neurometabolic and neurovascular coupling, and on cortical electrical activity, both in individuals with normal cognitive function and those affected by Mild cognitive Impairment and Alzheimer's Disease .

DETAILED DESCRIPTION:
Current pharmacological interventions mostly target symptoms. Most recently, disease-modifying therapies targeting beta-amyloid aggregation have been developed. Randomized controlled trials using these drugs (Lacenemab and Donanemab) in patients with early symptomatic AD showed a modest impact in terms of slowing cognitive decline and reducing amyloid biomarkers, associated with significant adverse effects. Yet, to date, no pharmacological intervention has been shown to reverse the loss in cognitive function associated with AD, nor to prevent the development of AD pathology. The risk of developing AD is influenced by both genetic and acquired factors, which include APOE genotype and insulin resistance. A better understanding of the association between insulin resistance and AD has important implications, both from a pathophysiological perspective and to foster the development of new therapeutic and preventive strategies. Observational studies have unambiguously demonstrated the bidirectional link between AD and type 2 diabetes mellitus (T2DM). Moreover, recent studies have shown that AD patients without T2DM have impaired insulin signalling at the brain level, which has led the field to define AD as "type 3 diabetes". Insulin is a hormone normally synthesized by the pancreas to regulate blood glucose levels and its utilization within the cells of our body, including the brain. To date, studies using intranasal insulin (INI) administration to investigate brain insulin signalling have shown significant variations in fMRI BOLD signal and improved cognition in healthy subjects. In AD patients, chronic INI administration for months showed that it significantly slowed down the progressive brain metabolism alteration as measured by positron emission tomography (PET) with 18-fluorodeoxyglucose (FDG), and to reduce the ratio of tau on amyloids deposit levels in cerebro-spinal fluid(tau-P181 to CSF Aβ42). Taken together, these findings raise the possibility that insulin is modifying AD-related processes.However, the effects of acute INI administration on brain function and cognition in healthy and AD subjects is not fully characterized yet. Acute INI could help to identify pathophysiologic processes occurring after a single doses, mainly insulin signalling and not due to any long term exposure event (genetic expression or modulation of the receptors).

PET-FDG is a neuroimaging technique that enables the quantification of human brain metabolism. Magnetic Resonance Imaging (MRI) utilizes a magnetic field to capture high-precision structural information about the humain brain. Functional MRI (fMRI) extends the capabilities of traditional MRI by capturing information on the modulation of brain perfusion during tasks and resting state. Finally, electroencephalography (EEG) allows direct and dynamic acquisition of cortical electric activity and allow to study functional brain connectivity.

Using simultaneous multimodal neuroimaging (FDG-PET, fMRI, EEG), this research project will aim to further investigate in vivo brain insulin signalling by exploring the effects of acute INI administration on neurometabolic and neurovascular coupling, and on cortical electrical activity, both in individuals with normal cognitive function and those affected by MCI/AD.

ELIGIBILITY:
Inclusion Criteria:

For the young subject group (group 1):

* Men and women aged 21-45 years old.
* Women under effective contraception.
* For Women, the study protocol should be performed during the follicular phase of the menstrual cycle, because of …
* Subjects must be proficient in speaking, reading and understanding French in order to be assessed with the neuropsychological tests battery.

For the MCI/AD group (group 2):

* Men and women aged 40-85 years old.
* Patients included on the registry of Neurodegeresence study in Hopital Erasme.
* Patients are capable of providing informed consent.
* Patients are proficient in speaking, reading and understanding French, in order to be assessed with the neuropsychological tests battery.
* Being diagnosed with amnestic MCI or probable mild AD, according to the core clinical criteria of the NIA and Alzheimer's Association guidelines.
* If the patient has a prescription medication acetylcholinesterase inhibitor (e.g. donepezil, rivastigmine, galantamine) and/or memantine doses has to be stable since 1 month at least.

For the group 2 - matched controls (group 3):

* Men and women aged 40-85 years old.
* Participants capable of providing informed consent
* Subjects are proficient in speaking, reading and understanding French, in order to be assessed with the neuropsychological tests battery.

Exclusion Criteria:

Exclusion criteria related to trimodal neuroimaging data acquisition:

* Dense or tight hair braiding or scalp lesions, preventing adequate EEG cap positioning.
* Pregnancy and/or breastfeeding.
* Claustrophobia.
* Metallic component (e.g. pacemaker) incompatible with the MRI acquisition.
* Participants over 120 kg for radioprotection issues.

Exclusion criteria related to demographic data:

* Any acute medical condition that required either hospitalization or surgery within the past 6 months.
* The subject has participated in a clinical trial investigation within 1 month of this study.
* Current or past psychiatric illness (according to the Mini International Neuropsychiatric Interview [MINI])
* For healthy participants (groups 1 and 3), having a first degree relative with dementia onset before 65 years (Alzheimer, Lewy body disease, Parkinson)
* Dementia (Mini-Mental State Examination [MMSE] scores ≤ 20) for group 2 and 3.
* CDR score ≥2, witch will be evaluated before inclusion by investigator for group 2 and 3.
* Current recreational drug or alcohol abuse.
* Serious systemic disease that would interfere with the conduction of the trial .
* Based on selection of Dementia from neurologic causes, Hachinski Ischemia Score > 4 (55).

Exclusion criteria related to the use of INI as IMP:

* Being under corticosteroid treatment (non-topical treatment)
* Being under birth-control pill containing ethinyl estradiol.
* The subject has an allergy to the IMP.
* History of bleeding disorder.
* The use of anticoagulants warfarin (Coumadin) or dabigatran (Pradaxa)
* Taking a hormonal therapy (e.g., post menopausal, oncological treatment…)
* Type 1 DM or Type 2 DM treated with insulin.
* History of severe hypoglycaemia.
* Participant being under any chronic Intranasal treatment.

Criteria susceptible to postpone study inclusion:

* Clogged or runny nose.
* Current Ears Nose Throat (ENT) infection.
* Fever during the last 24 hours.
* Consumption of caffeine during the last 24 hours.
* Fasting period inferior to 12h before study visits.
* Sleep deficiency the night preceding study days as assessed by Pittsburgh Survey

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Effects of INI administration on FMRI data in the 3 groups | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  For brain fRMI data: BOLD signal variation (Arbitrary Unit from a percent change from baseline).
Effects of INI administration on PET-FDG regional standardized data in the 3 groups | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  For brain PET-FDG: regional SUV value(standardized Uptake Ratio) .The SUV is a mathematically derived ratio of tissue radioactivity concentration at a point in time at a specific region of interest and the injected dose of radioactivity per kilogram of the patient's body weight
Effects of INI administration on PET-FDG global data in the 3 groups | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  For brain PET-FDG: Statistical Parametric Mapping analysis (SPM) for voxel-wise groups comparison and multiple correlations (t-score)
Effects of INI administration on EEG connectivity data in the 3 groups | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Connectivity changes (SmallWorldness index σ , a quantitative method for determining canonical network equivalence,)
Effects of INI administration on EEG Frequency band data in the 3 groups | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Spectrum analysis of the power (Power of the EEG signal(µV²/Hz) plotted against frequency band in Hz)

SECONDARY OUTCOMES:
Impact of gender on Intranasal insulin administration responses | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Co-analysis of primary endpoint: this variable will be included as covariable in group and population analysis (Male or Female)
Impact APOE (apolipoprotein E ) genetic status on Intranasal insulin administration responses | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Co-analysis of primary endpoint: this variable will be included as covariable in group and population analysis (Carrier , Homozygote , non-carrier)
Impact of Insulino-resistance scores ( Homeostatic Model Assessment of insulin resistance Scale (HOMA-IR) ), on Intranasal insulin administration responses | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Co-analysis of primary endpoint: this variable will be included as covariable in group and population analysis.
  higher Range of HOMA-IR indicate higher resistance to insulin. This scale is a ratio : Fasting glycaemia (mmol/L) * Fasting Insulinemia (mui/mL)/22.5.
  Cut off are defined with value <1.0 for non resistant subject. >1.9 for insulin resistance and >2.9 for high insulin resistance.
Impact of intranasal insulin administration on cognition and episodic memory | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Neuropsychological Data: A French-language battery for "Free Recall and Recall with Clue- 16" (RL-RI-16) The subjects get a global score from 0 to 144; a higher score means better-preserved memory function. Those score are then adjusted to existing data and deviation of the subject is calculated in statistical z-score.
Impact of intranasal insulin administration on attention / visual scanning | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Neuropsychological Data: Attention testing will be assessed with tests from a Attention Test Battery,validated in french, assessing the attention of the subject.
  Visual scanning a matrix-like arrangement of 5 x 5 stimuli is used, the aim being to detect whether this arrangement includes a critical stimulus or not. One reaction key is used for the answer "present" and another for the answer "not present".
  T Score are calculated for row and column , compared to a data base adjusted for age.
Impact of intranasal insulin administration on attention / mental flexibility | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Neuropsychological Data: This test is a "set shifting" task. A letter and a number are presented simultaneously to the right and left of the center of the screen. The subject has two reaction keys, one on the left and one on the right hand side. The task is to press the reaction key corresponding to the side on which the target stimulus appears.
  T Score are calculated from the reaction times, compared to a data base adjusted for age.
Impact of intranasal insulin administration on attention / inhibition. | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Neuropsychological Data: Attention testing will be assessed with tests from Attention Test Battery,validated in french, assessing the attention of the subject.
  Reaction times and errors are recorded in a simple Go/No-go test with two stimuli ""+"" and ""x"", of which only one (the ""x"") is critical
  T Score are calculated from reaction time, compared to a data base adjusted for age.
Impact of INI Administration on Spatial Memory | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Spatial memory testing will be assessed with the RUCHE-M test (Ruche Modified test).
  Scoring is 1 point for every square accurately reproduced in the learning phase; the same scoring will apply for the 5-time recall (total 50 points). For scoring the recognition test, 10/10 is attributed if the participant finds the correct grid. 1 point is subtracted for every failure.
  A lower score is attributed for lower performance in visual memory.
Impact of INI Administration on Global Memory Performance | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Score ranging from 0 to theoretically infinity, defined as how much a subject could memorize in serial information. A higher score means higher performance in sequential memory learning.
Impact of INI Administration on Fluency | end of acquisition for each group (each group of 30 subject estimated at 12 weeks after first subjet acquisition)
  Score goes from 0 to theoretically 120; the number of names a subject can present starting with the same letter.
  Performance is directly reflected in the score; higher scores report higher performances.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Leurquin-Sterk, MD,PhD, Principal Investigator — Nuclear Medicine department of H.U.B. site Erasme.; Xavier De Tiège, MD,PhD, Study Chair — Laboratoire de Neuroanatomie et Neuroimagerie translationnelles Université Libre de Bruxelles

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared on the CTIS database.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available Before the study start , being registered in CTIS database
Access Criteria: Publicly available
URL: https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en

REFERENCES:
- [Background] DeTure MA, Dickson DW. The neuropathological diagnosis of Alzheimer's disease. Mol Neurodegener. 2019 Aug 2;14(1):32. doi: 10.1186/s13024-019-0333-5. PMID 31375134
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Background] Dhana K, Aggarwal NT, Rajan KB, Barnes LL, Evans DA, Morris MC. Impact of the Apolipoprotein E epsilon4 Allele on the Relationship Between Healthy Lifestyle and Cognitive Decline: A Population-Based Study. Am J Epidemiol. 2021 Jul 1;190(7):1225-1233. doi: 10.1093/aje/kwab033. PMID 33585904
- [Background] Steen E, Terry BM, Rivera EJ, Cannon JL, Neely TR, Tavares R, Xu XJ, Wands JR, de la Monte SM. Impaired insulin and insulin-like growth factor expression and signaling mechanisms in Alzheimer's disease--is this type 3 diabetes? J Alzheimers Dis. 2005 Feb;7(1):63-80. doi: 10.3233/jad-2005-7107. PMID 15750215
- [Background] Tian S, Huang R, Han J, Cai R, Guo D, Lin H, Wang J, Wang S. Increased plasma Interleukin-1beta level is associated with memory deficits in type 2 diabetic patients with mild cognitive impairment. Psychoneuroendocrinology. 2018 Oct;96:148-154. doi: 10.1016/j.psyneuen.2018.06.014. Epub 2018 Jun 22. PMID 29957442
- [Background] Gudala K, Bansal D, Schifano F, Bhansali A. Diabetes mellitus and risk of dementia: A meta-analysis of prospective observational studies. J Diabetes Investig. 2013 Nov 27;4(6):640-50. doi: 10.1111/jdi.12087. Epub 2013 Apr 26. PMID 24843720
- [Background] Ott A, Stolk RP, van Harskamp F, Pols HA, Hofman A, Breteler MM. Diabetes mellitus and the risk of dementia: The Rotterdam Study. Neurology. 1999 Dec 10;53(9):1937-42. doi: 10.1212/wnl.53.9.1937. PMID 10599761
- [Background] de la Monte SM, Wands JR. Alzheimer's disease is type 3 diabetes-evidence reviewed. J Diabetes Sci Technol. 2008 Nov;2(6):1101-13. doi: 10.1177/193229680800200619. PMID 19885299
- [Background] Nijssen KMR, Mensink RP, Joris PJ. Effects of Intranasal Insulin Administration on Cerebral Blood Flow and Cognitive Performance in Adults: A Systematic Review of Randomized, Placebo-Controlled Intervention Studies. Neuroendocrinology. 2023;113(1):1-13. doi: 10.1159/000526717. Epub 2022 Aug 24. PMID 36219990
- [Background] Shpakov AO, Zorina II, Derkach KV. Hot Spots for the Use of Intranasal Insulin: Cerebral Ischemia, Brain Injury, Diabetes Mellitus, Endocrine Disorders and Postoperative Delirium. Int J Mol Sci. 2023 Feb 7;24(4):3278. doi: 10.3390/ijms24043278. PMID 36834685
- [Background] Wu S, Stogios N, Hahn M, Navagnanavel J, Emami Z, Chintoh A, Gerretsen P, Graff-Guerrero A, Rajji TK, Remington G, Agarwal SM. Outcomes and clinical implications of intranasal insulin on cognition in humans: A systematic review and meta-analysis. PLoS One. 2023 Jun 28;18(6):e0286887. doi: 10.1371/journal.pone.0286887. eCollection 2023. PMID 37379265
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Schmid V, Kullmann S, Gfrorer W, Hund V, Hallschmid M, Lipp HP, Haring HU, Preissl H, Fritsche A, Heni M. Safety of intranasal human insulin: A review. Diabetes Obes Metab. 2018 Jul;20(7):1563-1577. doi: 10.1111/dom.13279. Epub 2018 Apr 6. PMID 29508509
- [Background] Rosenbloom MH, Barclay TR, Pyle M, Owens BL, Cagan AB, Anderson CP, Frey WH 2nd, Hanson LR. A single-dose pilot trial of intranasal rapid-acting insulin in apolipoprotein E4 carriers with mild-moderate Alzheimer's disease. CNS Drugs. 2014 Dec;28(12):1185-9. doi: 10.1007/s40263-014-0214-y. PMID 25373630
- [Background] Hallschmid M. Intranasal Insulin for Alzheimer's Disease. CNS Drugs. 2021 Jan;35(1):21-37. doi: 10.1007/s40263-020-00781-x. Epub 2021 Jan 30. PMID 33515428
- See also: The Global Impact of Dementia: An analysis of prevalence, incidence, cost and trends — https://www.alzint.org/u/WorldAlzheimerReport2015.pdf